CLINICAL TRIAL: NCT03774953
Title: A Randomized, Controlled Clinical Trial on the Effect of Protein Supplement on Lean Body Mass in Patients With Community Acquired Pneumonia
Brief Title: The Effect of Protein Supplement on Lean Body Mass in Patients With Pneumonia
Acronym: CAPprotein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAP protein
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-08

CONDITIONS: Community-acquired Pneumonia
Keywords: pneumonia; community acquired pneumonia; protein; lean body mass; weight loss; readmission; infection
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia; Weight Loss; Infections | interventions — Proteins

STUDY DESIGN:
Intervention Model Description: Randomized to intervention or control arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): protein and vitamin supplementation
  Interventions: Dietary Supplement: Protein and vitamin supplementation
- Control group (No Intervention): No supplementations

INTERVENTIONS:
Dietary Supplement: Protein and vitamin supplementation — The intervention group will receive 1.5 g protein/kilo/day during hospitalization and a standard dose of 27 g protein/day in 60 days after discharged together with a daily dose of vitamin/mineral supplement
  Arms: Intervention group

SUMMARY:
The purpose of this clinical trial is to reduce the patient's loss of lean body mass by protein supplementation during hospitalization and 60 days after hospital discharge. Also, the study aims to reduce the risk of readmission to the hospital due to relapse or complications and thereby improving the overall health for the patients.

The intervention group will receive protein supplementation during hospitalization and after discharge, while the control group will continue their normal diet.

DETAILED DESCRIPTION:
Infections are globally the biggest cause of mortality. In Denmark community acquired pneumonia is one of the most common causes for infections in patients. Mortality in pneumonia has been stable high over the past 10 years. Therefore, it is relevant to look at improving the prognosis of these patients. After a longer period of hospitalization, patients generally have a poor condition with loss of body weight and lean body mass. Hereafter, patients must often undergo a longterm rehabilitation period and they become inactive and fatigue.

This is a threat for the patients, due to the fact that there is a higher risk of complications and readmissions.

Proteins are the body's building blocks. Thus, supplementing patients with a daily higher protein content, it is believed to reduce their loss of lean body mass, and thereby reduce the total loss of body weight as well. Protein supplementation together with vitamin- and mineral supplementation is thought to improve all these health risk markers for the patients.

Methods:

Inclusion: 40 men and women >60 years hospitalized with community acquired pneumonia Intervention: The patients will be randomized to either the control- or intervention group. They will receive the same treatment and care, the only difference is that the patients in the intervention group will receive protein- and vitamin supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with community acquired pneumonia
* >60 years
* Patients who are able to speak and understand Danish

Exclusion Criteria:

* Patients with hospitalized acquired pneumonia
* Patients with septic shock
* Patients with an active cancer and in cancer treatment
* Patients in dialysis
* ICU patients
* Patients unable or unwilling to give informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Loss of Lean Body Mass | Change from Baseline lean body mass until 2 months after discharged
  Loss of lean body mass measured by bioimpedance

SECONDARY OUTCOMES:
Loss of Body weight | Change from Baseline weight until 2 months after discharged
  Loss of body weight measured by weight scale
Readmissions | Up to 6 months
  Number of readmissions
Length of hospital stay between the two groups | From admission until discharge (an average of 5 days)
  Number of days
Quality of life measured by units on a scale | Change in individual experiences regards to quality of life from Baseline until 2 months after discharged
  Quality of life measured by units on a scale
Normal daily living function | Change in physical condition from Baseline until 2 months after discharged
  Normal daily living function measured by units on a scale

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte Lindegaard Madsen, Study Director — Nordsjaellands Hospital
Locations (1):
- Nordsjaellands hospital, Hillerød, Denmark